CLINICAL TRIAL: NCT06064786
Title: Evaluation of Fetuin-A and hsCRP Levels in Gingival Crevicular Fluid in Periodontitis Diabetic and Non-Diabetic Patients
Brief Title: Fetuin A Association in Periodontal Disease and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Tarrad, associate professor, Fayoum University
Other Study IDs: REC-FDBSU/03082023-2/ER
Record Dates: First submitted 2023-09-20; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — GCF samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 15 healthy patients with generalized periodontitis stage III.
  Interventions: Diagnostic Test: GCF levels of fetuin A and hsCRP evaluation
- Group II: 15 patients suffering from type 2 diabetes mellitus with generalized periodontitis stage III
  Interventions: Diagnostic Test: GCF levels of fetuin A and hsCRP evaluation
- Group III: 15 systemically healthy patients without periodontitis
  Interventions: Diagnostic Test: GCF levels of fetuin A and hsCRP evaluation

INTERVENTIONS:
Diagnostic Test: GCF levels of fetuin A and hsCRP evaluation — ELIZA kits are used for GCF levels of fetuin A and hsCRP evaluation

SUMMARY:
Aim: The aim of the current study was to compare and correlate gingival crevicular fluid (GCF) fetuin-A levels and high sensitivity C-reactive protein (hs-CRP) levels in non-diabetic periodontitis patients and type 2 diabetic periodontitis patients with healthy subjects and revealing its possible role in diagnosis of periodontal disease.

Methodology: Forty-five periodontitis stage III patients categorized into 3 groups according to whether having type II diabetes mellitus or not were compared to systemically and periodontally healthy participants in this investigation. Clinical parameters for all groups were recorded. Assessment of GCF levels of fetuin A and hs-CRP were done to all enrolled participants utilizing an enzyme linked immune-sorbent assay (ELISA) kit. Receiver operating characteristic (ROC) curve was performed to reveal sensitivity, specificity, predictive value and diagnostic accuracy of the markers used.

ELIGIBILITY:
Inclusion Criteria:

* both gender periodontitis stage III

Exclusion Criteria:

1. Smoking,
2. Systemic diseases (except DM in group B),
3. Periodontitis patients having periodontal treatment recently (past 6 months),
4. Pregnancy, lactation, contraceptive pills,
5. Anti-inflammatory/ immunosuppressive drugs.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: individuals recruited from outpatient clinic of periodontology department
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
GCF levels of fetuin A and hsCRP evaluation in all groups | levels of fetuin A and hsCRP are measured at baseline after the completion of all GCF sample collection carried at the day of enrollment of subjects in the investigation after diagnosis confirmation
  ELIZA kits

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No